CLINICAL TRIAL: NCT06932978
Title: The Impact of Smart Glasses on the Usability and Satisfaction of Operating an Environmental Control System or Communication Aid
Brief Title: The Use of Smart Glasses for Environmental Controls
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Lothian (Other Government)
Responsible Party: Principal Investigator, Graham Henderson, Chief Investigator, NHS Lothian
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: AC24008; 24/NW/0057 (Other: North West - Greater Manchester East Research Ethics Committee)
Record Dates: First submitted 2025-04-10; First posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Neurologic Disorder
Keywords: Environmental controls; Smart glasses; Activities of daily living; self-help devices; wearable technology
MeSH Terms: conditions — Nervous System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Smart glasses (Experimental): The participant will be provided with a set of smart glasses (X-REAL Air 2) as an alternative display for their existing environmental control system. They will have the smart glasses to trial for a period of 3 weeks.
  Interventions: Device: Provision of smart glasses for environmental control use

INTERVENTIONS:
Device: Provision of smart glasses for environmental control use — To the authors knowledge there has not been a clinical trial that includes the use of smart glasses with environmental controls. The smart glasses were used with environmental control systems that had a USB-C display output.

SUMMARY:
Environmental control systems are a type of assistive technology that can be controlled by a wide variety of different methods (e.g. switches) and can assist people with physical disabilities to control various electronic devices in the home. Communication aids are designed to assist people who have difficulties speaking to communicate. Both systems are designed to provide independence and potentially could have a positive effect on quality of life.

The majority of communication aid and environmental control systems aimed at high end users require a screen to be mounted in front of the user. The limitations with this are that the user is only able to access their device when it has been suitably mounted in front of them. There are occasions when mounting devices in front of the user is difficult due to other considerations for example transfers in and out of a wheelchair. As smart glasses can potentially be worn at all times during the day this could provide an effective alternative solution.

The purpose of this study is to explore with service users the usability and satisfaction provided by smart glasses when operating a communication aid/environmental control system. The study will achieve the above aim by undertaking a satisfaction questionnaire prior and post a 3 week trial of using smart glasses with their device. In addition an interview will be carried out with participants to explore the impact that smart glasses has had on the usability of their device.

Participants will be recruited by contacting eligible patients of the NHS Lothian Environmental Control Service and communication aid service. The end point of the study will be 8 months from the start date (allowing for follow up data to be collected for anyone recruited towards the end of the 6-month recruitment period).

ELIGIBILITY:
Inclusion Criteria:

* Existing environmental control system user (age 18-80).
* Neurological condition.
* Cognitive ability to answer the questions and to give consent.
* Current environmental control system is compatible with smart glasses display.

Exclusion Criteria:

* Current environmental control system or communication aid is not compatible with smart glasses display.
* Rapidly deteriorating condition

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2024-05-05 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Quest 2.0 | Baseline and 3 weeks
  This is a 12-item instrument that asks for the recipient to score their satisfaction of various aspects of an assistive technology device and service between 1 (not satisfied at all) and 5 (very satisfied). Eight of items relate to a device and four to the service, in this study due to the focus on the assistive technology device, only the answers relating to the device were collected. The instrument has been extensively used for assessing satisfaction with assistive technology and has been validated and tested for its reliability.

SECONDARY OUTCOMES:
Semi-structured interview | 3 weeks after provision of smart glasses
  The semi-structured interviews were conducted using six open-ended questions. The questions posed included ones relating to both satisfaction and usability. This included ones about the advantages, disadvantages and any points for improvement for the smart glasses. Additional questions included ones about making comparisons to using a traditional screen setup, how easy or hard the smart glasses were to use and whether participants would continue to use the smart glasses. When appropriate follow up questions were asked to elicit more information about answers.

CONTACTS AND LOCATIONS:
Locations (1):
- SMART Centre, Astley Ainslie Hospital, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Not required. A summary of the data in an anonymised form is sufficient.

DOCUMENTS (1):
  • Study Protocol (2024-03-07): https://cdn.clinicaltrials.gov/large-docs/78/NCT06932978/Prot_000.pdf